CLINICAL TRIAL: NCT07202741
Title: The Effect of Yoga on Pelvic Pain and Quality of Life in Women With Endometriosis
Brief Title: Effect of Yoga on Pelvic Pain and Quality of Life in Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gizem Cevik, PhD student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulUC-HEM-GÇ-01
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis
Keywords: Endometriosis; pelvic pain; quality of life; yoga
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: It is an experimental study consisting of 2 groups, a randomized controlled experiment and a control group, using a pre-test-post-test design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga group (Experimental): At the patient's first meeting, they were given an educational brochure and booklet about endometriosis and yoga. The researcher, who received an RYS-200 Yoga Instructor Certificate from the Turkish Yoga Federation, prepared a yoga video for endometriosis patients with a yoga instructor and shared it on Google Drive. The women practiced yoga according to the designated days and times. Yoga practiced three times a week for a total of eight weeks.
  Until the end of the 8th week, online yoga practices continued via Skype with the researcher twice a week and yoga practices that the participants would practice themselves once a week.
  Participants were encouraged to continue their yoga practice at least twice a week for the next four weeks with weekly motivational and follow-up messages. At the end of the 12 weeks, participants were contacted by phone to assess their yoga practice attendance and satisfaction, and they were asked to complete forms.
  Interventions: Other: yoga group
- control group (No Intervention): During the initial patient encounter, the researcher provided information about endometriosis, its symptoms, diagnosis, pain management methods, and ways to adopt a healthy lifestyle, all in a 20-minute session using a brochure and educational booklet. Participants were provided with a printed version of the educational booklet and brochure for later use.
  No intervention was administered for 8 weeks, and routine follow-up was conducted.
  At the end of weeks 4, 8, and 12, the Endometriosis Pain Monitoring Form, Visual Analog Scale (VAS), McGill Pain Scale Short Form, Endometriosis Health Profile Questionnaire (EHP-5), and Psychological Well-Being Scale were completed via telephone.

INTERVENTIONS:
Other: yoga group — A total of 50 minutes of hatha yoga practice was performed three times a week for 12 weeks.
  * In the first week, two days of face-to-face yoga practice with the researcher.
  * During the eighth week, online yoga practices were held twice a week via Skype with the researcher and one yoga practice per week (a list was made for the group the researcher would create via WhatsApp).
  The participants were supported with weekly motivation and follow-up information to continue practicing yoga at least twice a week for the next four weeks. All yoga sessions included a 10-minute warm-up and breathing session, 50 minutes of hatha yoga, 15 minutes of relaxation and separation, and 5 minutes of feedback. At the end of the session, the participants received support regarding correct yoga asanas, motivation, and consistency.
  Other Names: yoga
  Arms: yoga group

SUMMARY:
Women may experience loss of work/education and disruption in family relationships due to endometriosis-related symptoms. While surgical and medical treatments provide effective results in the management of endometriosis-related pain, the rate of recurrence is high. There is a need for nurse-led studies to identify supportive practices and interventions that can improve the quality of life and comfort of women with endometriosis, as well as to assess the effectiveness of these interventions. Nurses, with their holistic and patient-centered approach, play a crucial role. Therapeutic communication between nurses and patients during the diagnosis, treatment, and follow-up of endometriosis will contribute to disease management.

While there are limited studies worldwide examining the effects of yoga on pain and quality of life in women with endometriosis, no studies have been found in our country on the effectiveness of yoga on endometriosis. Therefore, this study was designed to contribute to the literature and evaluate the effects of yoga on pelvic pain and quality of life in women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 diagnosed with endometriosis
* Experiencing pelvic pain for at least 6 months (VAS score ≥4)
* Not pregnant
* Have not practiced yoga before
* Able to participate with internet access
* No communication barriers
* No health problems that would prevent practicing yoga
* No psychiatric health problems

Exclusion Criteria:

* Becoming pregnant during the study
* Developing a health problem that prevents yoga
* Failing to participate in at least two of the 8-week yoga program

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale for Pelvic Pain | 12 weeks
  The Visual Analog Scale is a widely used scale in daily practice to measure perceived pain. It consists of a measured horizontal or vertical line. A value of "0" indicates no pain on a 10 cm neck, a value of "1-4" indicates mild pain, "5-6" indicates moderate pain, and "7-10" indicates severe pain. A value of "10" indicates the most severe pain.
McGill Pain Scale Short Form for Pelvic Pain | 12 weeks
  The McGill Pain Scale Short Form consists of three sections. The first section contains 15 word groups describing the sensory/perceptual pain dimension (the first 11 words) and the emotional/emotional pain dimension (the last four words). Increasing total pain scores indicate an increase in the individual's perception of pain. The second section of the scale determines the severity of an individual's pain using a VAS. The third section uses a six-point Likert-type scale to determine the severity of the pain. The scale consists of expressive values ranging from 0 = no pain, 1 = mild, 2 = bothersome, 3 = distressing, 4 = excruciating, and 5 = unbearable pain. A low score indicates that the individual's pain intensity is generally low or mild, while a high score indicates high or severe pain.
Quality of life (Endometriosis Health Profile Questionnaire-5 score) | 12 weeks
  The Endometriosis Health Profile Questionnaire (EHP-5) consists of core (pain, control and powerlessness, emotional well-being, social support, and body image) and modular (work life, relationship with children, sexual life, healthcare professionals, treatment, and infertility) sections. Each item is scored on a four-point scale as 0, 1, 2, 3, and 4, corresponding to never, rarely, sometimes, often, and always. Scores are converted to a scale ranging from 0 to 100, representing best and worst health status, respectively. The total score on the scale increases as the quality of life improves.
Psychological well-being (Psychological Well-being Scale score) | 12 weeks
  The eight-item Psychological Well-Being Scale describes important elements of human functioning, from positive relationships and feelings of competence to having a meaningful and purposeful life. The scale's items are answered on a scale of 1-7, from strongly disagree (1) to strongly agree (7). All items are worded positively. Scores range from 8 (if all items are answered "strongly disagree") to 56 (if all items are answered "strongly agree"). A higher score indicates a higher level of psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: İlkay GÜNGÖR SATILMIŞ, Professor Dr., Principal Investigator — Florence Nightingale Faculty of Nursing, Department of Nursing, Department of Women's Health and Disease Nursing
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No